CLINICAL TRIAL: NCT02727192
Title: Sleep Disordered Breathing in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Effect of Treatment of Sleep Apnea in Patients With Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Health Association (Other); Medtronic (Industry); ResMed (Industry)
Responsible Party: Principal Investigator, Lars Gullestad, Professor MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gullestad
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Sleep Disordered Breathing; Sleep Apnea; Paroxysmal Atrial Fibrillation
Keywords: Atrial fibrillation; CPAP; Sleep apnea; Sleep disordered breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Atrial Fibrillation | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAP-therapy (CPAP or ASV) (Active Comparator): Patients are randomized to either intervention Group: Positive airway pressure therapy (PAP-therapy) or Control. Patients in the intervention arm will be treated with PAP-therapy (Continous Positive Airway Pressure (CPAP) or Adaptive Servo Ventilation (ASV).
  Interventions: Device: PAP (CPAP or ASV)
- Control group (No Intervention): No sleep apnea treatment

INTERVENTIONS:
Device: PAP (CPAP or ASV) — Patients will be randomized to treatment of Sleep Apnea with a CPAP or control
  Arms: PAP-therapy (CPAP or ASV)

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac rhythm disturbance in adults, with prevalence expected to rise significantly the coming decades. The occurrence of AF is associated with significantly increased mortality as well as morbidity of which cerebrovascular accidents is the most important. Unfortunately treatment options remain limited. Anti-arrhythmic drugs are widely used but have limited efficacy and the potential for toxicity and adverse events are recognized. Recent year's catheter ablation of AF continues to gain acceptance for symptomatic treatment, but recurrence rate are high with need for continuous medication. Thus there is a need to better understand what causes development and triggers episodes of AF as well to introduce new treatment options. Cardiometabolic factors such as obesity, inactivity and sleep apnea (SA) have therefore gained interest. Many patients with AF have chronic sleep apnea, and in the present study the investigators want to explore the interaction between SA and AF. The hypothesis of the present study is that SA may trigger AF and that treatment of SA will reduce the overall burden of AF as well as reduce the recurrence of AF after pulmonary vein ablation. To test the hypothesis the investigators will implant a Reveal device that continuously records the hearts rhythm of 100 patients with paroxysmal AF and concomitant SA. Initially the influence of SA on onset of AF will be examined, and the patients will then be randomized to treatment of SA or not and the influence on total AF burden recorded both before and after ablation.

DETAILED DESCRIPTION:
For the present project the investigators have established a research team from 2 different university hospitals. This team, including high ranked, internationally renowned scientist from both clinical and basic sciences, will make a framework for PhD candidates and will ensure the patient cohort. Patients with paroxysmal AF and SA will be examined with an extensive diagnostic battery including advanced cardiac imaging tools allowing a proper description of the heart. Then a Reveal that continuously monitor the rhythm of the heart will be inserted, allowing the influence of SA, physical activity, inflammatory parameters, and other external variables on total AF burden to be examined. The patients will then be randomized to treatment of SA with a CPAP or not, and the AF burden recorded 6 months before ablation and 6 months after.

The present investigations carried out, are expected to results in better understanding of the interaction between AF and SA and may lay the scientific basis for better diagnostic and therapeutic approaches for patients with AF. In addition, given the advantage of continuous Reveal® recording of the patient's heart rhythm, the present study will examine possible triggers of AF such as activity level and inflammatory substances, and examine the role of structural abnormalities in the heart as assessed by echocardiography for the triggering of AF episodes. An overall aim is therefore a better phenotyping of the patient which could aid in a more person-specific treatment approach, with direct consequences both for the individual patient and for the society.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Male or female
* Patients with paroxysmal AF scheduled for first or second catheter ablation
* Moderate-to-severe SA defined as an AHI ≥15/h (OSA and/or CSA)
* Signed informed consent

Exclusion Criteria:

* Unstable patients
* Patients with left ventricular ejection fraction (LV-EF) < 45%
* Unstable coronary artery disease, myocardial infarction or PCI within 3 months prior to the study
* Bypass surgery within 6 months prior to the study
* Patients with TIA or stroke within the previous 3 months
* BMI > 40kg/m2
* Drowsy drivers and/or sleepy patients with ESS (Epworth Sleepiness Score) > 15
* Patients with interstitial lung diseases, severe obstructive lung defects, and thoracic myopathies or severe obstructive lung defects with FEV1 < 50% of predicted
* Oxygen saturation < 90% at rest during the day
* Poor compliance
* Patients with single chamber pacemaker (or ICD)
* Current use of PAP therapy
* Patients using amiodarone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Traaen GM, Aakeroy L, Hunt TE, Overland B, Bendz C, Sande LO, Aakhus S, Fagerland MW, Steinshamn S, Anfinsen OG, Massey RJ, Broch K, Ueland T, Akre H, Loennechen JP, Gullestad L. Effect of Continuous Positive Airway Pressure on Arrhythmia in Atrial Fibrillation and Sleep Apnea: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2021 Sep 1;204(5):573-582. doi: 10.1164/rccm.202011-4133OC. PMID 33938787
- [Derived] Traaen GM, Aakeroy L, Hunt TE, Overland B, Lyseggen E, Aukrust P, Ueland T, Helle-Valle T, Steinshamn S, Edvardsen T, Khiabani Zare H, Aakhus S, Akre H, Anfinsen OG, Loennechen JP, Gullestad L. Treatment of sleep apnea in patients with paroxysmal atrial fibrillation: design and rationale of a randomized controlled trial. Scand Cardiovasc J. 2018 Dec;52(6):372-377. doi: 10.1080/14017431.2019.1567933. Epub 2019 Feb 5. PMID 30638392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 109 patients with paroxysmal atrial fibrillation and moderate to severe sleep apnea were included in the study and randomized to PAP-therapy or control. One patient refused further participation and was not included in the analysis. 108 patients were therefore included in the full set analysis.
  21 patients without sleep apnea or mild sleep apnea (AHI<15) were included as a reference group.
  Therefore, 130 patients were included in the study, but only 109 were included for randomization.
Pre-assignment Details: Before inclusion patients were invited to a CPAP mask tolerance test. Patients who complied with the treatment were invited to be included in the study.
  All patients were randomized to CPAP. In the CPAP group, one patient had CPAP treatment-emergent central SA shortly after randomization and was therefore switched to ASV.
Groups:
- CPAP-therapy: CPAP-therapy (Continous Positive Airway Pressure)
- Control Group: No sleep apnea treatment (usual care)
- ASV-therapy: ASV-therapy (Adaptive Servo-Ventilation)
Period: Overall Study
Arm/Group | CPAP-therapy | Control Group | ASV-therapy
Started | 54 | 54 | 1
Completed | 53 | 54 | 1
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PAP-therapy (CPAP or ASV): PAP-therapy (Continous Positive Airway Pressure (CPAP) or Adaptive Servo Ventilation (ASV).
- Total: Total of all reporting groups
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.4) | 62.1 (7.8) | 62.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 39 | 43 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 54 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Norway | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change in AF Burden
Description: Difference between PAP treatment and usual care in change of AF burden (% of time in AF, as measured by loop recorder) from baseline (one month prior to randomization) to the last three months of the five month intervention period.
Time Frame: Baseline (pre-randomization) was the first month of loop recorder data collection and was compared to the last three months of the intervention period.
Measure: Mean (Standard Deviation); unit: percentage of time in AF
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
percentage of time in AF
  Baseline | 5.6 (8.3) | 5.0 (8.9)
  Last three months of intervention | 4.1 (6.5) | 4.3 (9.4)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.520, Regression, Linear — A two-sided significance level of 5% was considered to indicate statistical significance; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.6 to 1.3]

2. Secondary Outcome: Change in AF Burden
Description: Difference between PAP treatment and usual care in change of AF burden (% of time in AF, as measured by loop recorder) from baseline (one month prior to randomization) to the last month of the intervention period.
Time Frame: Baseline to the last month of intervention period
Measure: Mean (Standard Deviation); unit: percentage of time in AF
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
percentage of time in AF
  Baseline | 5.6 (8.3) | 5.0 (8.9)
  Last month of the intervention period | 4.6 (8.1) | 5.1 (10.8)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.440, Regression, Linear; Mean Difference (Net) = -0.9, 95% CI 2-sided [-3.3 to 1.5]

3. Secondary Outcome: Change in AF Burden
Description: Difference between PAP treatment and usual care in change of AF burden (% of time in AF, as measured by loop recorder) from baseline (one month prior to randomization) to the last five months of the intervention period (the whole intervention period).
Time Frame: Comparing Baseline to the last five months of the intervention period
Measure: Mean (Standard Deviation); unit: percentage of time in AF
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
percentage of time in AF
  Baseline | 5.6 (8.3) | 5.0 (8.9)
  5 months intervention period | 4.5 (6.4) | 4.6 (9.8)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.410, Regression, Linear; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.1 to 0.9]

4. Secondary Outcome: Number of Participants With More Than 25% Reduction in AF Burden
Description: Difference between PAP treatment and usual care in the proportion of patients with at least 25% reduction of AF burden (% of time in AF, as measured by loop recorder) from baseline (one month prior to randomization) to the last three months of the intervention period.
Time Frame: Baseline to last three months of the intervention
Population: The proportion of patients with at least 25% reduction in AF burden
Measure: Count of Participants; unit: Participants
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
Participants | 22 | 17
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.33, Chi-squared; Difference in Percentage of Participants = -9.3

5. Secondary Outcome: Change of Recurrence Rate After Ablation, as Measured by Loop Recorder
Description: Change of recurrence rate after ablation, as measured by loop recorder, after 6 months post ablation and after 12 months post ablation.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2021-12

6. Secondary Outcome: Change in AF Symptoms as Assessed by Atrial Fibrillation Severity Scale (AFSS)
Description: Change in AF symptoms between CPAP treatment and usual care. The questionnaire quantifies three domains of AF: event frequency (score 1-10), duration (score 1-10), and global episode severity (score 1-10). The total AF burden is calculated from the modified sum of the frequency, duration, and severity of AF (score 3-30, with higher scores indicating greater AF burden ). In addition, the AFSS assesses a symptom score based on seven items asking how bothered patients are by specified symptoms (score 0-35). Global well-being is a visual analogue scale ranging from 1 to 10 (10 indicating the best possible life).
Time Frame: 6 months, 12 months and 18 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Quality of Life (QoL) as Assessed by Medical Outcomes Study 36-item Short-Form Health Survey (SF-36)
Description: Difference between CPAP and usual care in QoL as assessed by SF36, Version 1.2. Item scores are transformed into the Physical and Mental Component Summary scores (PCS and MCS). Scores range from 0 to 100, with higher scores indicating a better health state.
Time Frame: Assessed at baseline, 6 months, 12 months and 18 months, baseline and 6 months reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale
  Baseline Mental Component Summary score | 49.9 (9.5) | 52.8 (6.6)
  Follow up 6 months Mental Component Summary score | 52.5 (8.7) | 51.5 (8.8)
  Baseline Physical Component Summary score | 43.1 (9.1) | 43.3 (10.2)
  Follow up 6 months Physical Component Summary score | 43.6 (10.2) | 45.9 (9.6)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Mental Component Summary score; Test type: Superiority; p = 0.058, Regression, Linear; Mean Difference (Net) = 2.8, 95% CI 2-sided [-0.1 to 5.8]
Statistical Analysis 2: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Physical Component Summary score; Test type: Superiority; p = 0.160, Regression, Linear; Mean Difference (Net) = -2.1, 95% CI 2-sided [-5.1 to 0.8]

8. Secondary Outcome: Change in Sleep Quality and Symptoms of Sleep Apnea: Epworth Sleepiness Scale (ESS) Score
Description: Difference between PAP treatment and usual care in Change in daytime sleepiness as measured using the Epworth Sleepiness Scale (ESS) score, with scores ranging from 0 to 24 (most sleepy)
Time Frame: 6 months, 12 months and 18 months. Baseline and 6 months reported
Population: Baseline and 6 months reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale
  Baseline | 8.2 (3.1) | 7.5 (3.3)
  Follow up 6 months | 7.1 (3.6) | 7.5 (3.7)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.110, Regression, Linear; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.0 to 0.2]

9. Secondary Outcome: Change in Symptoms of Obstructive Sleep Apnea Assessed by the Berlin Questionnaire.
Description: Change in sleep quality and symptoms of obstructive sleep apnea as measured using the Berlin Questionnaire. Positive scores in two or more categories suggest a high risk of OSA.
Time Frame: 6 months, 12 months and 18 months
Reporting Status: Not Posted, anticipated posting 2022-12

10. Secondary Outcome: Change in Symptoms of Sleep Apnea Using the Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: Change in sleep quality and symptoms of obstructive sleep apnea as measured using the Functional Outcomes of Sleep Questionnaire (FOSQ). Score range is 5-20 Points, with higher scores indicating better functional status.
Time Frame: 6 months, 12 months and 18 months. Baseline and 6 months reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
score on a scale
  Baseline | 17.4 (1.9) | 17.7 (2.0)
  Follow up 6 months | 17.6 (2.0) | 17.7 (2.0)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.850, Regression, Linear; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.6]

11. Secondary Outcome: Change in Symptoms of Sleep Apnea Measured by the STOP-Bang
Description: Change in sleep quality and symptoms of obstructive sleep apnea as measured using the STOP-Bang Questionnaire. Score between 0-8. A score of ≥3 suggest risk for OSA.
Time Frame: 6 months, 12 months and 18 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in CRP
Description: Difference between PAP treatment and usual care in change of CRP
Time Frame: 6 months, 12 months and 18 months. Baseline and 6 months reported.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
mg/L
  Baseline | 1.2 [0.8 to 1.9] | 1.0 [0.8 to 2.6]
  Follow up 6 months | 1.0 [0.7 to 2.1] | 1.1 [0.8 to 2.3]
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.650, Regression, Linear; Median Difference (Net) = 0.3, 95% CI 2-sided [-1.0 to 1.6]

13. Secondary Outcome: Change in Left Ventricular Ejection Fraction
Description: Difference between PAP treatment and usual care in change of left ventricular ejection fraction as assessed by ecco
Time Frame: 6 months, 12 months and 18 months. Baseline and 6 months reported.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
percentage
  Baseline | 58.5 (5.2) | 57.9 (5.2)
  Follw up 6 months | 59.4 (4.2) | 56.6 (5.2)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.006, Regression, Linear; Mean Difference (Net) = 2.6, 95% CI 2-sided [0.8 to 4.5]

14. Secondary Outcome: Change in the Cardiac Marker NT-proBNP.
Description: Difference between PAP treatment and usual care in change of Cardiac marker of NT-proBNP.
Time Frame: 6 months, 12 months. Baseline and 6 months reported.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
ng/L
  Baseline | 95.5 [50 to 152.3] | 84 [50 to 170.5]
  Follow up 6 months | 102.5 [50.7 to 190.3] | 87 [50 to 229.5]
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.389, Regression, Linear; Median Difference (Net) = -31.4, 95% CI 2-sided [-103.4 to 40.7]

15. Secondary Outcome: Examine the Effect of SA Treatment on Gene Expression of White Blood Cells.
Description: Examine the effect of SA treatment on gene Expression of white blood cells. Is paroxysmal AF Associated with specific gene Expression patterns? Examine the influence of SA treatment on the pattern of gene Expression and if this is related to reduction of atrial fibrillation burden
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

16. Secondary Outcome: Examine if Onset of Paroxysmal AF is Associated With Specific Activity Patterns, as Assessed by Garmin Vivofit2/3, Activity Recording
Description: Examine if onset of paroxysmal AF is Associated with specific Activity patterns, as assessed by garmin Vivofit2/3, Activity recording
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

17. Secondary Outcome: Change in Body Composition as Assessed by Bioelectric Impedance Analysis (BIA) (Tanita)
Description: Change in body composition (BMI) as assessed by Bioelectric Impedance Analysis (BIA) (Tanita)
Time Frame: Baseline to follow up 6 months
Measure: Mean (Standard Deviation); unit: Kg/m ̂ 2
Arm/Group | PAP-therapy (CPAP or ASV) | Control Group
Number analyzed (Participants) | 54 | 54
Kg/m ̂ 2
  Baseline | 29.8 (4.8) | 29.8 (4.1)
  Follow up 6 months | 29.6 (5.1) | 29.6 (4.2)
Statistical Analysis 1: Comparison: PAP-therapy (CPAP or ASV) vs Control Group; Test type: Superiority; p = 0.697, Regression, Logistic; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.5]

18. Secondary Outcome: Lung Function Test as Assessed by Spirometry
Description: Lung function test as assessed by spirometry
Time Frame: Baseline, 6 months
Reporting Status: Not Posted, anticipated posting 2022-12

ADVERSE EVENTS:
Time Frame: 5 months (intervention period)
Description: Adverse event collection was obtained by regular investigator assessment, and data collection from the loop recorder (prolonged pauses).
Groups:
- CPAP-therapy: Positive airway pressure therapy (CPAP)
- ASV Therapy: Adaptive Servo Ventilation (ASV)
Arm/Group | CPAP-therapy | Control Group | ASV Therapy
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/53 | 2/54 | 0/1
Other Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP-therapy (N=53) | Control Group (N=54) | ASV Therapy (N=1)
Pacemaker implantation due to syncope and prolonged pauses (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Hospitalization due to syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization due to symptomatic atrial fibrillation (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0)
Hospitalization due to chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization due to hemorrhagic stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT02727192/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT02727192/SAP_000.pdf